CLINICAL TRIAL: NCT00158639
Title: Electronic Communications and Home Blood Pressure Monitoring
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01HL075263 (NIH); R01 HL075263-01A1-01
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Hypertension
Keywords: Blood Pressure Monitoring, home; Pharmaceutical services; Self care
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Home BP;secure messaging;pharmaceutical care;

SUMMARY:
The control of blood pressure (BP) for patients with hypertension on medications has been elusive, despite the availability of evidence-based nationally recognized guidelines for treatment and 30 years of research addressing this. At present, less than 50% of patients with known hypertension are adequately controlled. If BP control could be improved, significant decreases in cardiovascular morbidity and mortality would occur.

The purpose of this study is to conduct a randomized controlled trial of the effectiveness of the provision of home blood pressure measurement and electronic communications (secure messaging to health care providers) to improve hypertension control.

DETAILED DESCRIPTION:
This is single-blind, randomized, controlled trial, to test the effectiveness of applying the chronic care model to hypertension.

There is an emerging consensus that multifaceted, multilevel, interventions are most effective in improving care for chronic conditions. In order to successfully plan and execute the required strategies, care planning is being increasingly conducted by the use of systems planning models. Since its original description by Wagner, Austin and Von Korff in 1996, the Chronic Care Model has found wide application, acceptance and success in planning care for chronic diseases, however to our knowledge, it has not yet been applied to the care of hypertension. There are six components of the model, including: clinical information systems, decision support, delivery system design, self-management support, organizational support, and community resources. The model describes these components to activate both patients and physicians, and when this occurs optimally, health outcomes improve. The interventions below are designed according to this construct and to determine whether enhanced patient self-management support in the form of home blood pressure monitoring and augmented delivery system design with pharmaceutical care improves hypertension control.

* Group-1 (Usual Care) will receive usual care for their hypertension. This includes the following for physicians: guidelines and decision support for treatment of hypertension, reminds and feedback as to medication choices, the use of electronic medical records with the ability to graphically display blood pressures over time. Patients have access to secure Intranet services already available at GHC including portions of their electronic medical record (including their blood pressures and the graphic display of these), messaging, and prescription refill services, and laboratory results.
* Group-2 (Blood Pressure Monitoring) will additionally receive home blood pressure monitors, instruction on their use, and a proficiency training session on Web-based communication and encouraged to use this to communicate their blood pressures with their physician, refill medications, and view parts of their medical records (blood pressures, labs, medication list).
* Group-3 (Blood Pressure Monitoring and Pharmaceutical Care) will receive all of the above plus planned and proactive, self and care management support provided by clinical pharmacists via the Web. One of three clinical pharmacists will be assigned to each patient in group 3. The clinical pharmacist will initially telephone the patient and do an intake visit to assess their medical history specific to hypertension care and assist the patient in designing an action plan that addresses blood pressure self-monitoring, medication use, lifestyle habits to reduce blood pressure and cardiovascular risk (they will assist the patient in choosing one lifestyle activity to work on), and follow-up plans. The pharmacist and patient will communicate at regular intervals by secure message (telephone and clinic visits will be occur if needed) and work collaboratively to improve blood pressure control. The pharmacist will use a medication algorithm (based on Group Health and JNC7 guidelines) to adjust medications until goal blood pressure is reached (<135 mmHg and <85 mmHg average for home BP measurements) and will provide information as to resources available within Group Health or the community to assist patients with their lifestyle goals. Record keeping will occur in the electronic medical record with key aspects shared electronically and securely with the patient and their physician.

The interventions will be delivered over a period of 12-months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hypertension in the prior two years and on hypertension medications
* Access to the Internet and an e-mail address
* Ability to use a computer using the English language
* Medical care coverage which permits them to refill prescriptions at Group Health Cooperative pharmacies and a willingness to do so.
* Blood pressure on each of two screening visits averaging > 90 mmHg diastolic or > 140 mmHg systolic and < 110 mmHg diastolic or < 200 mmHg systolic

Exclusion Criteria:

* Diagnosed or history of diabetes, cardiovascular disease (ischemic heart disease, valvular heart disease, heart failure, arrhythmias, strokes or transient ischemic attacks, and peripheral vascular disease)
* Current treatment for cancer, on immunosuppressant or antiretroviral treatment.
* Surgery or hospitalization in the prior 3 months
* Pregnancy (or plans to become pregnant in the next 12 months)
* Plans to move out of the area or leave the health plan in the next 12 months.
* Upper arm circumference size > 18 inches.
* Arrhythmia detected at screening visits

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 778 (Actual)
Dates: Start 2005-06; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
*change in mean diastolic, systolic, and combined diastolic and systolic BP.
*percent of patients with adequately controlled BP.

SECONDARY OUTCOMES:
*adherence to recommended anti-hypertensive medications and the proportion on preferred anti-hypertensive medications.
*patients' general health status, sense of self-efficacy in their management of hypertension, and satisfaction with their care in general and that for hypertension.
*to assess the impacts of each intervention on hypertension visits, primary care visits, and medication use for hypertension, and estimate the incremental cost-effectiveness of each.

CONTACTS AND LOCATIONS:
Overall Officials: Beverly B Green, MD, MPH, Principal Investigator — Kaiser Permanente
Locations (1):
- Group Health Research Institute, Seattle, Washington, United States

REFERENCES:
- [Derived] Meenan RT, Anderson ML, Chubak J, Vernon SW, Fuller S, Wang CY, Green BB. An economic evaluation of colorectal cancer screening in primary care practice. Am J Prev Med. 2015 Jun;48(6):714-21. doi: 10.1016/j.amepre.2014.12.016. PMID 25998922
- [Derived] Green BB, Anderson ML, Ralston JD, Catz SL, Cook AJ. Blood pressure 1 year after completion of web-based pharmacist care. JAMA Intern Med. 2013 Jul 8;173(13):1250-2. doi: 10.1001/jamainternmed.2013.1037. No abstract available. PMID 23689927
- [Derived] Green BB, Anderson ML, Ralston JD, Catz S, Fishman PA, Cook AJ. Patient ability and willingness to participate in a web-based intervention to improve hypertension control. J Med Internet Res. 2011 Jan 20;13(1):e1. doi: 10.2196/jmir.1625. PMID 21371993
- [Derived] Green BB, Cook AJ, Ralston JD, Fishman PA, Catz SL, Carlson J, Carrell D, Tyll L, Larson EB, Thompson RS. Effectiveness of home blood pressure monitoring, Web communication, and pharmacist care on hypertension control: a randomized controlled trial. JAMA. 2008 Jun 25;299(24):2857-67. doi: 10.1001/jama.299.24.2857. PMID 18577730